CLINICAL TRIAL: NCT03043287
Title: Voiding Efficiency, a Predictor of CIC
Brief Title: Voiding Efficiency, a Predictor of Clean Intermittent Catheterization (CIC)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: CMO-US-URO-0506
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BOTOX®: Participants who received 100 to 200 units (U) onabotulinumtoxinA (BOTOX®) as treatment for OAB. No study drug is administered in this study.
  Interventions: Biological: onabotulinumtoxinA

INTERVENTIONS:
Biological: onabotulinumtoxinA — onabotulinumtoxinA (BOTOX®)100 to 200 U
  Other Names: Botulinum Toxin Type A; BOTOX®

SUMMARY:
This study is a retrospective chart review of patients treated with onabotulinumtoxinA (BOTOX®) for idiopathic overactive bladder (OAB) and will determine voiding efficiency (VE) cutoff ratios that predict post-procedure urinary retention requiring catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Patient with documented idiopathic OAB diagnosis
* Patient was treated with 100-200U of BOTOX® for OAB
* Urodynamics assessment within prior to first BOTOX® injection.

Exclusion Criteria:

* Patient had received botulinum toxin formulations other than BOTOX® in the bladder
* Patient had symptoms of OAB associated with a neurological condition (eg, spinal cord injury, multiple sclerosis, cerebrovascular accident, Alzheimer's disease, Parkinson's disease, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with BOTOX® for Idiopathic OAB in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Pre-BOTOX® Injection VE Cutoff-Ratios that Predict the Risk of CIC following Treatment with 100-200U of BOTOX® | Pre-BOTOX® Injection (Baseline)
  VE was calculated as the ratio of voided volume to the total bladder capacity.
Length of Time of CIC Use in Clinical Practice after Treatment with 100-200U BOTOX® | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dana Fetterolf, Study Director — Allergan
Locations (3):
- United States (3):
  - Regional Urology, Shreveport, Louisiana
  - Chesapeake Urology Associates, LLC, Baltimore, Maryland
  - Virginia Urology, Richmond, Virginia

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com